CLINICAL TRIAL: NCT00313417
Title: A Double-blind, Parallel, Randomized, add-on Clinical Trial of Creatine Versus Placebo Added to Antidepressant Treatment of Patients With Major Depressive Episode.
Brief Title: Creatine as a New Therapeutic Strategy in Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Herzog Hospital (Other)
Collaborators: Beersheva Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Levine Yossi Prof., HEAD OF PSYCHIATRIC WARD, Herzog Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Shapira1CTIL
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Major Depressive Disorder
Keywords: Creatine; major depressive disorders
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: Creatine monohydrate
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — Up to 10 grams
  Arms: 1
Other: Placebo — Placebo will be given in the same way and appearance as the active treatment
  Arms: 2

SUMMARY:
Creatine as a new therapeutic strategy in depression:

A double-blind, parallel, randomized, add-on clinical trial of creatine versus placebo added to antidepressant treatment of patients with major depressive episode.

DETAILED DESCRIPTION:
Dr.Boris Nemetz and Prof.Joseph Levine M.D., Beer Sheva Mental Health Center,Israel.

Creatine plays a pivotal role in brain energy homeostasis, being a temporal and spatial buffer for cytosolic and mitochondrial pools of the cellular energy currency adenosine triphosphate (Wyss & Kaddurah-Daouk, 2000). Recent studies have suggested increased brain utilization of oxygen following oral creatine supplementation (Persky & Brazeua, 2001). Creatine supplementation is widely used in enhancing sports performance, and has been tried in the treatment of neurological, neuromuscular and atherosclerotic disease with a paucity of side effects (Persky & Brazeua, 2001).

Creatine enters the brain via a specialized sodium dependent transporter. Dechent et al (1999) studied the effect of oral creatine supplementation of 20g/day for 4 wk demonstrating a significant increase of mean concentration of total creatine across brain regions (8.7% corresponding to 0.6mM, P < 0.001). Lyoo et al (2003) studied magnetic resonance spectroscopy of high-energy phosphate metabolites in human brain following oral supplementation of creatine reporting that creatine (0.3 g/kg/day for the first 7 days and 0.03 g/kg/day for the next 7 days) significantly increased brain creatine levels.

Accumulated evidence suggests the possible involvement of altered cerebral energy metabolism in the pathophysiology of depression (Mayberg, 1994). Functional brain imaging studies (positron and single photon emission tomography) have shown decreased blood flow and metabolism in the frontal lobes and basal ganglia in unipolar depression (Kennedy et al, 2001; Derevets et al, 2002).

Proton magnetic resonance spectroscopy studies have studied brain levels of creatine-containing compounds. Kato et al (1992) reported that phosphocreatine was significantly decreased in severely (as opposed to mildly) depressed patients. Dager et al (2004) studied depressed or mixed-state bipolar patients using two-dimensional proton echo-planar spectroscopic imaging, reporting an inverse correlation between severity of depression and white matter creatine levels.

Finally, several studies suggest that agents with reported antidepressant activity may increase brain levels of creatine containing compounds. Sartorius et al (2003) used MRS to study metabolic changes in the hippocampus of rats and demonstrated a significant creatine level rise induced by electroconvulsive shock treatment occurring specifically in the group of animals which had exhibited depression-like [learned helplessness] behaviour before the ECT.

S-adenosyl-L-methionine (SAM) and acetyl-L-carnitine - both reported to have antidepressant effects - have increased brain phosphocreatine levels in healthy subjects (Silveri et al, 2003) and in geriatric depressed patients (Pettegrew et al, 2002) respectively.

Taken together, these findings suggest the possibility of using oral creatine supplementation to increase brain levels of creatine containing compounds and therefore, most likely by modifying high-energy phosphate metabolism in hypoactive brain areas, to treat subjects with major depression.

Open study of creatine in depression: A preliminary open study of creatine monohydrate (Roitman S, Green T, Osher Y, Karni N and Joseph Levine, submitted), suggested a statistically significant beneficial effect of creatine augmentation to antidepressant treatment in resistant major depression, but possible precipitation of a manic switch in resistant bipolar depression (see table 1 for results). Adverse reactions were mild and transitory and included mild nausea and flatus.

Ww propose to perform a double-blind, parallel, randomized add-on clinical trial of creatine versus placebo added to current antidepressant treatment in the treatment of major depressive disorder in the early phase of treatment resistant major depressive episode.

Early phase of treatment resistant depressive episode is defined where the current treatment resistant depressive episode lasts no more than 6 months.

Based on the results of the open study presented in Tab.1, we hypothesize that such study will show a statistically significant and clinically relevant difference between the active treatment (creatine) and placebo in the double blind add-on trial design proposed below.

Study design

This study is a parallel, randomized, double blind, placebo controlled, 4 weeks clinical trial examining the effect of creatine versus placebo added to antidepressant treatment of subjects with major depression demonstrating lack of adequate response to the current antidepressant treatment, administered in adequate dose for at least 3 weeks.

Creatine will be purchased from Solgar LTD, Israel, where 1 tablet contains 1 gram.

Forty consenting patients, women and men, 18 - 75 years old will be recruited. All subjects will have a primary diagnosis of major depression, and at the time of recruitment will be experiencing a major depressive episode with a duration ≥ 3 weeks and < 6 months. Subjects will be eligible to enter the study only if they will have a minimum score of 18 points on the 24-item Hamilton Rating Scale for Depression (HAMD) and are receiving conventional antidepressant treatment in adequate dose for at least 3 weeks with no more than mild improvement Blood cell count, liver and kidney functions will be performed before entering the study, only in patients who have not had them performed during the last 6 month prior to entering the study.

Pregnant or lactating patients, those with clinically significant or unstable medical conditions, epilepsy, or a history of alcohol or substance abuse will be excluded from this study. All participants will be monitored weekly and will have a 24 hours telephone access to the researcher, and those who will develop suicidal or aggressive behaviors that may endanger themselves or others, will be immediately discontinued from the study.

The researcher evaluating the HAM-D as well as the other study scales will be blind to the add-on treatment (creatine or placebo). Twenty patients will be treated with creatine add-on for 4 weeks (up to 10 grams).

The other 20 patients will be receiving placebo add-on for 4 weeks. Patient's antidepressant treatment will not be changed during the study participation.

Benzodiazepines are allowed, but the dose will not exceed Lorazepam equivalent dose of 4 mg daily.

The following data will be recorded at the beginning of the study:

Demographic data Psychosocial data History of hospitalizations Comorbid medical conditions Family history of affective disorders Previous pharmacological treatments and treatment response Seasonal pattern of depressive symptomatology

The following scales will be completed at the beginning of the study and weekly thereafter (weeks 1 to 4):

Hamilton Depression Rating Scale (24 items) Clinical Global Impression Backwards digit span test Scale for the assessment of side effects

The main outcome measure will be the prediction of a sustained ≥ 50 % decrease of the Hamilton Depression Scale (HAM-D) total score versus baseline ('sustained response') and the presence of ≥20 % HAM-D total score improvement after 1 weeks of treatment('early improvement')and the presence of ≥50 % HAM-D total score improvement after 1 weeks of treatment ('very early improvement') .

References

Wyss M, Kaddurah- Daouk R. Creatine and creatinine metabolism. Physiol Rev 2000; 80: 1107-213.

Persky AM, Brazeau GA. Clinical pharmacology of the dietary supplement creatine monohydrate.

Pharmac Rev 2001; 53: 161-76.

Dechent P., Pouwels PJ. Wilken B. et al. Increase of total creatine in human brain after oral supplementation of creatine-monohydrate.

Am J Physiol 1999; 277. R698-798.

Lyoo IK, Kong SW, Hirashima F. et al. Multinuclear magnetic resonance spectroscopy of high-energy phosphate metabolites in human brain following oral supplementation of creatine- monohydrate.

Psychiatry Res 2003; 123:87-100.

Mayberg HS. Frontal lobe dysfunction in secondary depression. J Neuropsychiatry Clin Neuroscience 1994; 6:428-442.

Kennedy SH, Evans KR, Kruger S, Mayberg HS, Meyer JH, McCann S, Arifuzzman AI, Houle S, Vaccarino FJ. Changes in regional brain glucose metabolism measured with positron emission tomography after paroxetine treatment of major depression.

Am J Psychiatry 2001 Jun;158(6):899-905.

Drevets WC, Bogers W, Raichle ME. Functional anatomical correlates of antidepressant drug treatment assessed using PET measures of regional glucose metabolism.

Eur Neuropsychopharmacol 2002 Dec;12(6):527-44.

Kato T, Takahashi S, Shioiri T, Inubushi T: Brain phosphorous metabolism in depressive disorders detected by phosphorus-31 magnetic resonance spectroscopy. J Affect Disord 1992; 26(4):223-30.

Dager SR, Friedman SD, Parow A, Demopulos C, Stoll AL, Lyoo IK, Dunner DL, Renshaw PF: Brain metabolic alterations in medication-free patients with bipolar disorder.

Arch Gen Psychiatry 2004; 61(5):450-8.

Sartorius A, Vollmayr B, Neumann-Haefelin C, Ende G, Hoehn M, Henn FA: Specific creatine rise in learned helplessness induced by electroconvulsive shock treatment.

Neuroreport 2003; 14(17):2199-2200.

Silveri MM, Parow AM, Villafuerte RA, Damico KE, Goren J, Stoll AL, Cohen BM, Renshaw PF: S-adenosyl-L-methionine: effects on brain bioenergetic status and transverse relaxation time in healthy subjects.

Biol Psychiatry 2003; 54(8):833-9.

Pettegrew JW, Levine J, Gershon S, Stanley JA, Servan-Schreiber D, Panchalingam K, McClure RJ: 31P-MRS study of acetyl-L-carnitine treatment in geriatric depression: preliminary results.

Bipolar Disord 2002; 4(1):61-6.

ELIGIBILITY:
Inclusion Criteria:

Age:18-75 -

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale, CGI | 4 weeks of treatment for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Levine, Prof., Principal Investigator — Beer Sheva Mental Health Center Israel.; Boris Nemets, Dr., Principal Investigator — Beer Sheva Mental Health Center Israel.
Locations (1):
- Beer Sheva Mental Health Center, Beersheba, Israel